CLINICAL TRIAL: NCT06898437
Title: Clinical Trial to Evaluate the Antitumor Efficacy and Safety of 177Lu-LNC1004 Injection in Patients With Fibroblast Activating Protein (FAP)-Positive Radioiodine-refractory Differentiated Thyroid Cancer (RAIR-DTC) Who Have Failed TKIs Treatment or Refuse Standard Treatment
Brief Title: Study of 177Lu-LNC1004 Injection in FAP-positive Radioiodine-refractory Differentiated Thyroid Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yansong Lin, Prof. M.D, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K7531
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Radioiodine Refractory Differentiated Thyroid Cancer
Keywords: Thyroid cancer; 177Lu-LNC1004; FAP
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-LNC1004 Injection (Experimental): All subjects will be administered with 177Lu-LNC1004 Injection at 80 mCi per cycle for 2 cycles with interval of 6 weeks.
  Interventions: Drug: 177Lu-LNC1004 Injection

INTERVENTIONS:
Drug: 177Lu-LNC1004 Injection — Intravenous administration: a single dose of 80 mCi per Cycle

SUMMARY:
177Lu-LNC1004 Injection, a radiopharmaceutical targeting FAP, has demonstrated preliminary antitumor effect in advanced FAP-positive solid tumor patients. The primary purpose of this study is to evaluate the efficacy of 177Lu-LNC1004 Injection in patients with FAP-positive RAIR-DTC who have failed first-line TKIs treatment or refuse standard treatment. All subjects will receive 80 mCi (± 10%) 177Lu-LNC1004 Injection intravenously every 6 weeks for 2 cycles.

DETAILED DESCRIPTION:
This prospective, single-arm, open label, single-center clinical trial is planned to enroll approximately 20 RAIR-DTC subjects s who have failed TKIs treatment or refuse standard treatment. All subjects will receive 80 mCi (± 10%) 177Lu-LNC1004 Injection intravenously every 6 weeks for 2 cycles. Disease progression and occurrence of AEs will be monitored during the trial. Based on tumor response assessment and AEs occurrence in the first 2 cycles, subjects may continue to receive 177Lu-LNC1004 Injection for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have the ability to understand and sign an approved informed consent form (ICF).
2. Aged 18 years or older, regardless of sex.
3. Histologically or cytologically confirmed RAIR-DTC subject who has failed TKIs treatment or refuse standard therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
5. At least one measurable lesion as defined by Response Criteria in Solid Tumors (RECIST) version 1.1.
6. Life expectancy of at least 6 months.
7. FAP-positive lesion confirmed by FAPI PET/CT scan.
8. Adequate organ function as defined by：

   * Bone marrow function: hemoglobin ≥ 100 g/L, neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L;
   * Liver function: albumin ≥ 3.0 g/dL; total bilirubin ≤ 1.5 × ULN; ALT and AST < 3 × ULN without liver metastasis or < 5 × ULN with liver metastasis;
   * Renal function: creatinine clearance ≥ 60 mL/min.
9. Clinically significant toxic reactions related to prior antitumor treatment that have recovered to Grade ≤ 1 (CTCAE V5.0).

Exclusion Criteria:

1. Known central nervous system metastases, except for the following:

   * Subject without clinical symptoms can be included in this trial after evaluation by the investigator.
   * Brain metastases that have been previously treated and confirmed by image to be stable for at least 4 weeks.
2. Secondary malignancy was detected within 5 years prior to first dosing, excluding cured localized carcinoma including cervical carcinoma in situ, basal cell skin cancer, and prostate cancer in situ, etc.
3. Received antitumor treatment including chemotherapy, radiotherapy, immunotherapy, and traditional Chinese medicine, etc. within 4 weeks prior to first dosing.
4. Subject who previously received targeted therapy, but discontinued treatment for less than 4 weeks or 10 half-lives prior to first dosing.
5. Received systemic radionuclide therapy or radioembolization within 6 months before first dosing or any external beam radiotherapy within 2 weeks before the first dosing.
6. Known allergy to 177Lu-LNC1004 Injection or similar drugs.
7. Subject has not fully recovered from major surgery prior to first dosing or expects to have major surgery during the study period.
8. Accompanied with severe cardiovascular and cerebrovascular diseases, including but not limited to:

   * Subject who has undergone coronary angioplasty, coronary stent placement, coronary artery bypass grafting, or implantation of defibrillation devices due to arrhythmia within 6 months;
   * There are serious heart rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block, etc.
   * Clinically significant abnormal ECG during the screening period, including QTcF > 470 ms in male and QTcF > 480 ms in female.
   * New York College of Cardiology (NYHA) grade ≥ 3.
   * Aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular event (NCI CTCAE v5.0) within 6 months.
9. Subject who has active and clinically significant bacterial, fungal, viral infection, or any other uncontrolled active infections such as active tuberculosis within 4 weeks prior to first dosing.
10. Known human immunodeficiency virus (HIV) infection or positive HIV test, positive syphilis antibody test, or active hepatitis except for:

    * Subject who is positive for hepatitis B surface antigen can be enrolled if HBV DNA level is less than 1×104 copies/mL or 2000 IU/mL, and can receive antiviral treatment according to clinical judgment during the trial.
    * Subject who is positive for HCV antibodies can be enrolled if HCV RNA test is negative.
11. Previously received allogeneic hematopoietic stem cell transplantation or organ transplantation.
12. Subject who has pleural effusion or ascites that required treatment or is deemed uncontrollable by investigator.
13. Subject who has mental illness or substance abuse, which may affect adherence to the trial.
14. Subject who refuses to take effective contraceptive measures during sexual intercourse from ICF signing to 6 months after last investigational drug administration；
15. Women who are pregnant or breastfeeding, or planning to become pregnant during the study period or within 6 months after last investigational drug administration；
16. Any other medical condition, metabolic abnormality, physical abnormality, laboratory abnormality, or other condition that the investigator deems inappropriate for study participation, or that would affect the interpretation of the study results, or place the subject at high risk, such as idiopathic pulmonary fibrosis or lung disease, urinary incontinence, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 24 months
  ORR is defined as the the proportion of subjects who achieve a best overall response of Complete Response (CR) or Partial Response (PR).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 24 months
  DCR is defined as the proportion of subjects who achieve a best overall response of CR, PR or Stable Disease (SD).
Duration of Response (DoR) | up to 24 months
  DoR is defined as the time from the earliest date of documented CR or PR until documented disease progression or death, whichever occurs first.
Progression Free Survival (PFS) | up to 24 months
  PFS is defined as the time from the first dose of 177Lu-LNC1004 Injection to the date of documented disease progression or death, whichever occurs first.
Biochemical Response (BR) | up to 24 months
  BR is defined as the percentage of change in serum Thyroglobulin (Tg) from baseline.
Safety | up to 24 months
  Adverse Event (AE), Serious Adverse Event (SAE), Treatment related Adverse Event (TRAE).

CONTACTS AND LOCATIONS:
Overall Officials: Peking Union Medical College Hospital, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China